CLINICAL TRIAL: NCT04988191
Title: The Efficacy and Safety of Toripalimab Combined With Bevacizumab and Chemotherapy as Neoadjuvant Therapy in Patients With Advanced MSI-H or dMMR Colorectal Cancer: an Open-label, Multicenter, Single-arm, Phase Ib/II Study
Brief Title: Toripalimab Plus Bevacizumab and Chemotherapy as Neoadjuvant Therapy in Advanced MSI-H or dMMR Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-115
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined with bevacizumab and chemotherapy (Experimental)
  Interventions: Drug: Toripalimab; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Toripalimab — Neoadjuvant therapy: Toripalimab is given by intravenous infusion at 3mg/kg d1 every 2 weeks for 3 cycles.
  Adjuvant therapy: Toripalimab is given by intravenous infusion at a dose of 240mg every 3 weeks for up to 9 cycles.
Drug: Bevacizumab — Neoadjuvant therapy: Bevacizumab is given by intravenous infusion at 5mg/kg d1 every 2 weeks for 3 cycles.
Drug: Irinotecan — Neoadjuvant therapy: Irinotecan is given by intravenous infusion at 180mg/m2 d1 every 2 weeks for 2 cycles.

SUMMARY:
This is a trial investigating the efficacy and safety of Toripalimab combined with bevacizumab and chemotherapy as neoadjuvant therapy in patients with advanced microsatellite instability-high (MSI-H) or DNA mismatch repair-deficient (dMMR) colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma meeting any of the following criterion: a) T3-4 resectable rectal cancer; b) T1-2 rectal cancer located within 12 cm from the anal verge and refusing direct surgery or radiation therapy; c) T4a-b resectable colon cancer.
2. Microsatellite instability-high (MSI-H) or DNA mismatch repair-deficient (dMMR).
3. Measurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria and haven't received any local treatment.
4. Eastern Cooperative Oncology Group (ECOG) 0-1.
5. Fully aware of this study and having signed informed consent.
6. Age 18 to 75 years old without gender limitation.
7. Good compliance.
8. Absolute neutrophil count ≥1500/mm3, platelet ≥100,000/mm3, Hb ≥10g/dl, serum creatinine ≤1.5 times ULN, creatinine clearance rate ≥50mL/min, ALT and AST ≤2.5 times ULN, INR or aPTT ≤1.5 times ULN (INR ≤2 times ULN and aPTT in normal range for patients who are on prophylactic anticoagulant therapy within 14 days before study treatment), total bilirubin level ≤2 times ULN (within 7 days before study treatment).
9. Women of childbearing age should confirm that serum pregnancy test is negative and agree to use effective contraceptive methods during study treatment and the following 60 days.

Exclusion Criteria:

1. Previously received anti-PD1 or anti-PDL1 or anti-PDL2 or anti-CTLA4.
2. Uncontrolled active bleeding from the primary tumor or intestinal obstruction.
3. Contraindications of bevacizumab or irinotecan.
4. Hypersensitivity to other monoclonal antibodies.
5. Any active, known or suspected autoimmune disease.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites to a moderate or greater extent.
7. History of one of the following dieases: idiopathic pulmonary fibrosis, organized pneumonia (eg. bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia and interstitial pneumonia, or evidence of active pneumonia through enhanced chest CT screening.
8. Major surgery within 4 weeks before enrollment and haven't fully recovered from the previous surgery.
9. Active bleeding or abnormal coagulation (aPTT >43s or INR >1.5 times ULN), or having a tendency to bleed or receiving thrombolytic or anticoagulant therapy.
10. Previously received allogeneic stem cell or parenchymal organ transplantation.
11. Any significant clinical or laboratory abnormality that the investigator considers to influence the safety assessment, eg. uncontrolled active infection, uncontrolled diabetes, hypertension that cannot be reduced to normal range with monotherapy, grade II or above peripheral neuropathy, congestive heart failure, heart disease (class II or higher) as defined by the New York College of Cardiology, myocardial infarction within 3 months prior to enrollment, unstable arrhythmias, unstable angina pectinis, chronic kidney disease, abnormal thyroid function and previous or co-existing malignancies.
12. History of uncorrected serum electrolyte disturbances such as potassium, calcium and magnesium.
13. HIV infection.
14. Active hepatitis B or hepatitis C.
15. Pregnancy or lactation period, or unwilling to use contraception during the trial.
16. With other malignancy within 5 year, except cervical carcinoma in situ, basal or squamous skin cancer, local prostatic carcinoma and ductal carcinoma in situ.
17. Use corticosteroids (dose of prednisone or similar drugs> 10mg/day) or other immunosuppressive agents within 14 days before enrollment.
18. Patients with active tuberculosis (TB) who are receiving anti-TB treatment or have received anti-TB treatment within 1 year.
19. Active infection, or treatment with oral or intravenous antibiotics within the first 2 weeks prior to neoadjuvant therapy, except prophylactic administration.
20. Anti-infective vaccine (eg. influenza vaccine, varicella vaccine, etc.) injection within 4 weeks before neoadjuvant therapy.
21. Previous participation in other clinical trials within 4 weeks before neoadjuvant therapy.
22. Any other disease, metabolic disorder, abnormal physical examination or abnormal laboratory results that may contrainn the use of trial drug, or affect the reliability of study results, or lead to high risk of treatment complications, or affect patient compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-06-24 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate based on blinded, independent, central review | 10 weeks
  Percentage of patients who achieve pathological complete response (pCR) based on blinded, independent, central review (BICR).

SECONDARY OUTCOMES:
R0 recession rate | 10 weeks
  Percentage of patients who achieve R0 recession.
Time to surgery | 10 weeks
  Measure of time from study treatment to surgery.
Pathological complete response rate assessed by local investigator | 10 weeks
  Percentage of patients who achieve pathological complete response (pCR) based on assessment of local investigator.
Pathological complete response rate based on blinded, independent, central review (BICR) and the assessment of local investigator | 10 weeks
  Percentage of patients who achieve pathological complete response (pCR) based on both blinded, independent, central review (BICR) and assessment of local investigator.
Tumor regression grade (TRG) | 10 weeks
Objective response rate | Up to 3 years
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).
Event free survival | Up to 3 years
  Measure of time from study treatment to disease progression or death.
Disease-free survival | Up to 3 years
  Measure of time from the date of surgery to disease relapse or death.
One-year or two-year disease-free survival rate | Up to 2 years
  Percentage of patients who achieve disease-free survival lasting for more than one and two years respectively from the date of surgery.
One-year or two-year overall survival rate | Up to 2 years
  Percentage of patients who achieve survival for more than one and two years respectively from date of first dose.
Score of life quality | Until 30 days after the last treatment
  Accessment of life quality based on EORTC QLQ-C30 and EORTC QLQ-CR29 scale.
Incidence of Treatment-Related Adverse Events | Until 30 days after the last treatment
  Number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Z, Wang X, Zhang X, Leng J, Cui M, Zhang J, Wang Q, Sun Y, Xu T, Chen M, Li J, Shen L. Toripalimab, bevacizumab, and irinotecan in dMMR/MSI locally advanced colorectal cancer: First-stage results from a phase 1b/2 trial. Cell Rep Med. 2025 Sep 16;6(9):102296. doi: 10.1016/j.xcrm.2025.102296. Epub 2025 Aug 15. PMID 40818457